CLINICAL TRIAL: NCT01931917
Title: A Randomised Controlled Pilot Trial of The Incredible Years Parents and Babies Program in Denmark
Brief Title: The Incredible Years Parents and Babies Program in Denmark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SFI 2570
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Parenting
Keywords: Prevention; Parenting; Infants; Family programs; Early intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IY Parents and Babies Program (Experimental): In the Incredible Years Parents and Babies Program, parents learn how to help their babies feel loved, safe, and secure. They learn how to encourage their babies' physical and language development. The parenting group format fosters peer support networks and shared learning. Trained Incredible Years facilitators use video clips of real-life situational vignettes to support the training and stimulate parenting group discussions and practice exercises with their babies. The program is group based with 6-8 mothers and partners attending 8 2 hour sessions with their babies.
  Interventions: Behavioral: Incredible Years Parents and Babies Program
- Usual Care (Active Comparator): Usual care consists of the elements that are being offered to all mothers in the participating municipalities which is 5 home visits by health visitors, a mothers group, a health nurse station and extra visits if needed.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Incredible Years Parents and Babies Program — 4-5 home visits by health visitor IY parents and babies program 8 sessions Group of mothers Health visitor station Extra visits by health visitor if needed
  Arms: IY Parents and Babies Program
Behavioral: Usual Care — 4-5 home visits by health visitor Group of mothers Health visitor station Extra visits by health visitor if needed
  Arms: Usual Care

SUMMARY:
The purpose of the pilot study is to examine the effects of the Incredible Years Baby Programme (IY baby) offered as a universal intervention compared to Usual Care (UC) for parents with infants aged 0-12 months.

DETAILED DESCRIPTION:
A randomised controlled effectiveness pilot trial of the Incredible Years Parents and Babies Program (IY baby)offered as a universal intervention in two municipalities in Denmark. 120 families will be randomised to IY Baby (intervention) og Usual Care (UC- control). Families recruited to the study have infants aged 0-4 months old. All first time mothers in one municipality and all mothers in another municipality are recruited. Outcomes are measured at 20 weeks post baseline and when the child is 18 months old. The aim of this trial is to estimate the effectiveness of the IY Baby program on parent and infant well-being, development and relationship and establish parameters for a definitive trial. In addition, the pilot study will also gather information on parent recruitment and participation to inform future research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Parents with a child aged 0-4 months
* Parents are able to understand Danish at a basic level

Exclusion Criteria:

* Serious physical disability
* serious mental disability
* Child can not be placed in out of home care

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Karitane Parenting Confidence Scale (KPCS) | Baseline, 20 weeks post intervention start
  The KPCS measures perceived parenting self-efficacy (PPSE) in parents of children aged 0-12 months. High PPSE has been shown to act as a buffer against factors that can compromise a child's development, such as parental depression, anxiety, stress and relationship difficulties, and is associated with actual parenting competence and positive child outcomes
  The KPCS is a short self-report instrument. It was developed in Australia primarily for health professionals experienced in working with parentcraft and psychosocial issues of early parenthood, including Maternal, Child and Family Health Nurses, and allied health and medical professionals.
Parental Stress Scale (PSS) | 20 weeks post intervention start, child age 18 months

SECONDARY OUTCOMES:
Sense of coherence (SOC13) | Baseline
Major Depression Inventory (MDI) | Baseline, 20 weeks post intervention start, child age 18 months
Ages and stages - Social-Emotional (ASQ-SE) | Baseline, 20 weeks post intervention start, child age 18 months
World health organisation well being index (WHO5) | Baseline, 20 weeks post intervention start, child age 18 months
Rosenberg self esteem (RSS) | 20 weeks post intervention start
Emotional Availability Scales (EAS) or Care Index | 20 weeks post intervention start
  Video observation task measuring mother-infant attachment and relation
Mother and baby interaction scale (MABISC) | 20 weeks post intervention start
Strengths and Difficulties Questionnaire (SDQ) | child age 18 months
Cognitive development questionnaire (CDQ) | child age 18 months
Being a Mother (BaM13) | child age 18 months
Parental Reflective Functioning Questionnaire (PRFQ-1) short version | child age 18 months
Parenting Sense of Competence (PSOC) | child age 18 months

OTHER OUTCOMES:
Parent and child health | 20 weeks post intervention start, child age 18 months
  Single items on parent and child health, child temperament, parent life satisfaction, network, economy, interaction with child, child height and weight.
Single items on child temperament | Baseline, 20 weeks post intervention start, child age 18 months
Single items on interaction with child | 20 weeks post intervention start, child age 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maiken Pontoppidan, Principal Investigator — VIVE - The Danish Center for Social Science Research
Locations (1):
- SFI the Danish National Centre for Social Research, Copenhagen, Denmark

REFERENCES:
- [Derived] Pontoppidan M, Thorsager M, Steenhoff T. Parent-child Relationship Outcomes of the Incredible Years Parents and Babies Program: A Pilot Randomized Controlled Trial. Scand J Child Adolesc Psychiatr Psychol. 2022 Jun 7;10(1):40-52. doi: 10.2478/sjcapp-2022-0004. eCollection 2022 Jan. PMID 35799975
- [Derived] Pontoppidan M, Klest SK, Sandoy TM. The Incredible Years Parents and Babies Program: A Pilot Randomized Controlled Trial. PLoS One. 2016 Dec 14;11(12):e0167592. doi: 10.1371/journal.pone.0167592. eCollection 2016. PMID 27974857
- [Derived] Pontoppidan M. The effectiveness of the Incredible Years Parents and Babies Program as a universal prevention intervention for parents of infants in Denmark: study protocol for a pilot randomized controlled trial. Trials. 2015 Sep 2;16:386. doi: 10.1186/s13063-015-0859-y. PMID 26329163
- See also: Paper - post intervention outcomes — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0167592
- See also: Trial protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-015-0859-y